CLINICAL TRIAL: NCT07239843
Title: Synapsing's Multinational Sociodemographic Study
Brief Title: Prospective Observational Study of the Relationship Between Sociodemographic Factors, Blood-based Biomarkers and Psychiatric Symptoms in Neurodegenerative Diseases and Mental Disorders
Acronym: Synapsing-SD
Status: Enrolling by invitation | Type: Observational
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Collaborators: University of Ulm (Other); University Of Perugia (Other); University of Eastern Finland (Other); Martin-Luther-Universität Halle-Wittenberg (Other)
Responsible Party: Sponsor
Other Study IDs: IIBSP-EPM-2024-176
Record Dates: First submitted 2025-11-14; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-08

CONDITIONS: Major Depressive Disorder (MDD); Schizophenia Disorder; Bipolar 1 Disorder; Alzheimer Disease; Parkinson Disease; Frontotemporal Dementia (FTD); Dementia With Lewy Bodies (DLB)
Keywords: magnetic resonance imaging; sociodemographic; biomarker; plasma; serum; blood
MeSH Terms: conditions — Depressive Disorder, Major; Alzheimer Disease; Parkinson Disease; Frontotemporal Dementia; Lewy Body Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Biospecimen Retention: Samples With DNA — Blood (plasma, serum)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- major depressive disorder: Clinical diagnosis of major depressive disorder
- Bipolar disorder: Clinical diagnosis of type I + II Bipolar disorder
- Schizophrenia: Clinical diagnosis of schizophrenia
- Parkinson's disease: Clinical diagnosis of Parkinson's disease
- Alzheimer's disease: Clinical diagnosis of Alzheimer's disease
- Dementia with Lewy bodies: Clinical diagnosis of dementia with Lewy bodies
- Unaffected controls: No clinical diagnosis of a primary psychiatric disorder or neurodegenerative disease

SUMMARY:
This is a prospective observational study to identify sociodemographic factors that predict mental health outcomes in the European population and provide evidence linking common, modifiable sociodemographic risk factors for psychiatric symptoms with biological changes in patients suffering from a mental disorder (MD) or a neurodegenerative disease (ND).

DETAILED DESCRIPTION:
Sociodemographic studies in mental disorder (MD) and neurodegenerative diseases (ND). Sociodemographic factors increase the likelihood of developing an MD and contribute to poorer outcomes. There is less research on socioeconomic differences in ND, but also low socioeconomic status is also associated with dementia risk and early onset dementia. Substantial gaps remain in understanding the social and biological mechanisms underlying these disparities. Effective public health interventions to reduce the burden of these disorders are currently lacking.

ELIGIBILITY:
Inclusion Criteria:

* Age>18 and donation of blood,
* full clinical and psychological assessment
* Available neuroimaging is optional as not all patients are suitable.
* Age and sex-matched unaffected volunteers without a MD or ND diagnosis are used as controls.
* Unaffected controls are usually spouses or children of patients that are informed about our studies at each clinical site.

Exclusion Criteria:

* Lack of neuropsychological data,
* anticoagulant treatment such as acenocoumarol, heparin, warfarin, dabigatran, rivaroxaban, apixaban, drug abuse in the last year,
* medical history of cancer affecting the central nervous system that has not been in complete remission for 5 years or longer,
* the patient has received potentially neurotoxic chemotherapy and/or patient has received cranial radiotherapy.
* Clinical diagnosis of Alzheimer's disease where pathophysiological markers (measured in CSF or plasma) are inconsistent with Alzheimer's disease pathophysiology.
* Cognitively healthy volunteers where pathophysiological markers (measured in CSF or plasma) are consistent with Alzheimer's disease or other neurodegenerative pathophysiology.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from specialized clinics at Barcelona (Spain), Perugia (Italy), Ulm (Germany), Halle (Germany) and Kuopio (Finland). Target % female in schizophrenia (30%), major depressive disorder (50%), bipolar disorder and controls (55%), Alzheimer's disease and controls (60%), frontotemporal dementia (65%), controls (65%). These percentages match those typically found in these disorders. Unaffected controls are usually spouses or children of patients that are informed about our studies at each clinical site. This study also includes participants from a wider European population of people with a lived experience of mental health issues from six focus countries of Europe, UK, Spain, Germany, Finland, Italy and Ireland.
Sampling Method: Non-Probability Sample
Enrollment: 1310 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2029-12-30 (Estimated)

PRIMARY OUTCOMES:
Diagnosis | 2-months after enrollment
  Primary diagnosis following evaluation by clinician and neuropsychologist or information relating to a previous or current MD/ND diagnosis or mental health issue (Anxiety disorders, behavioural and emotional disorder in children, bipolar affective disorders, depression, dissociation and dissociative disorders, eating disorders, obsessive compulsive disorder, paranoia, post-traumatic stress disorder or psychosis).
Perceived Wellbeing and Mental Health | 2-months after enrollment
  Total Score on the Perceived Wellbeing and Mental Health section of the survey
Social support | 2-months after enrolment
  Total score on the Social support section of the sociodemographic survey
Socioeconomic background | 2-months after enrollment
  Total score on the Socioeconomic background section of the sociodemographic survey
Health behaviour | 2-months after enrollment
  Total score on the Health behaviour section of the sociodemographic survey
Hamilton Depression Rating Scale | 2-months after enrollment
  Total score on the Hamilton Depression Rating Scale
Boston Naming Test | 2-months after enrollment
  Total score on the Boston Naming Test

SECONDARY OUTCOMES:
Structural brain changes | 2 months after enrollment
  Acquisition of 3T-MRI with a high-resolution 3D T1-weighted anatomical image, a multi-shell diffusion-weighted MRI, and a resting-state functional sequence.
Synaptic biomarker | Blood extracted 2-months after enrollment
  Plasma concentration of (e.g., NPTX2) measured in plasma

CONTACTS AND LOCATIONS:
Locations (1):
- IRSP, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No